CLINICAL TRIAL: NCT00002718
Title: A Phase II Trial of T-Cell Depleted Marrow Grafts Combined With Infusions of G-CSF Stimulated, CD34 Ceprate Stem Cell Column Selected, E-Rosette Depleted Peripheral Blood Progenitor Cells Derived From HLA Haplotype Matched Related Donors for Patients With Leukemia Lacking an HLA-Matched Related or Unrelated Donor
Brief Title: T-cell Depleted Bone Marrow and G-CSF Stimulated Peripheral Stem Cell Transplantation From Related Donors in Treating Patients With Leukemia, Lymphoblastic Lymphoma, Myelodysplastic Syndrome, or Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95-084; P30CA008748 (NIH); MSKCC-95084; NCI-V96-0809
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood acute lymphoblastic leukemia; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; stage IV adult lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; juvenile myelomonocytic leukemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; chronic myelomonocytic leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic | interventions — Antilymphocyte Serum; Filgrastim; Cyclophosphamide; Cytarabine; Methylprednisolone; Thiotepa; Radiotherapy

ARMS (1):
- Candidates for transplant (Experimental): Pts stratified by number of HLA-incompatible alleles(1 vs 2 or 3). Harvest:Begin 6-10 d before transplant,allogeneic BM is harvest & tx in vitro. Begin 5-6 d before transplant,G-CSF-stimulated,PBSC harvest,selected for CD34+ cells,& treatment in vitro. If doable,ABM harvest in event of allogeneic graft failure. Myeloablation:Pts u/g TBI 3x d days -9 to -6, thiotepa IV over 4hrs days -5 & -4, & cyclophosphamide IV days -3 & -2. Transplant:CD34+, E-rosette & T-cell-depleted PBSC infuse over 15mins & T-cell-depleted bone marrow infused over 1-5mins day 0. Pts get G-CSF IV over 30 min begin day 1 & continue til blood counts recover & tapering. Pts get anti-thymocyte globulin IV over 4-6hrs days 8,10,12,&14 & oral methylprednisolone days 8-14 followed by tapered doses days 15-17. See detailed description for more details.
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: methylprednisolone; Drug: thiotepa; Procedure: in vitro-treated bone marrow transplantation; Procedure: in vitro-treated peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Drug: cyclophosphamide
Drug: cytarabine
Drug: methylprednisolone
Drug: thiotepa
Procedure: in vitro-treated bone marrow transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow and peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of T-cell depleted bone marrow and G-CSF stimulated peripheral stem cell transplantation in treating patients with leukemia, lymphoblastic lymphoma, myelodysplastic syndrome, or aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the potential of T-cell-depleted bone marrow and peripheral blood stem cells (PBSC) from HLA-haplotype, partially matched related donors to induce extended disease-free survival in patients with leukemia, lymphoblastic lymphoma, myelodysplastic syndrome, or severe aplastic anemia who would otherwise be ineligible for transplantation because of the lack of an HLA-identical related or unrelated donor.
* Determine the impact of filgrastim (G-CSF)-stimulated, CD34+, E-rosette and T-cell-depleted PBSC derived from an HLA-haplotype, partially matched donor on the incidence and quality of engraftment, kinetics, and quality of hematopoietic and immunologic reconstitution, and incidence and severity of graft-versus-host disease (GVHD) in these patients.
* Correlate the doses of PBSC and clonable T-cells with the incidence of engraftment, extent of chimerism, incidence and severity of acute and chronic GVHD, characteristics of hematopoietic and immunologic reconstitution, and overall and disease-free survival rates at 2-4 years after transplantation in these patients.

OUTLINE: Patients are stratified by number of HLA-incompatible alleles (1 vs 2 or 3).

* Harvest: Beginning 6-10 days before transplantation, allogeneic bone marrow is harvested and treated in vitro. Beginning 5-6 days before transplantation, filgrastim (G-CSF)-stimulated, allogeneic peripheral blood stem cells (PBSC) are harvested, selected for CD34+ cells, and treated in vitro. If feasible, autologous bone marrow is harvested in the event of allogeneic graft failure.
* Myeloablation: Patients undergo total body irradiation 3 times a day on days -9 to -6, thiotepa IV over 4 hours on days -5 and -4, and cyclophosphamide IV on days -3 and -2.
* Transplantation: CD34+, E-rosette and T-cell-depleted PBSC are infused over 15 minutes and then T-cell-depleted bone marrow is infused over 1-5 minutes on day 0. Patients receive G-CSF IV over 30 minutes beginning on day 1 and continuing until blood counts recover and then tapering. Patients receive anti-thymocyte globulin IV over 4-6 hours on days 8, 10, 12, and 14 and oral methylprednisolone on days 8-14 followed by tapered doses on days 15-17.
* CNS prophylaxis: Beginning at least 2 months after transplantation, patients with acute lymphocytic leukemia (ALL) and no history of CNS leukemia receive cytarabine intrathecally (IT) monthly for 6 months and patients with ALL and a history of CNS leukemia receive cytarabine IT monthly for 12 months.

Patients with graft failure are offered autologous bone marrow transplantation (BMT) or second allogeneic BMT.

Patients are followed at 1, 3, 6, and 12 months and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Acute myelogenous leukemia (AML) meeting 1 of the following conditions:

    * Failed to achieve first remission after an intensive induction regimen containing an anthracycline and cytarabine
    * In second remission and not enrolled in a protocol for autologous bone marrow transplantation
    * Failed to achieve or sustain second remission
    * In first remission but at high risk of relapse because of 1 of the following factors:

      * High-risk cytogenetic features (monosomy 7,5q-, trisomy 8, or t(9;22))
      * AML secondary to treatment of a prior malignancy and without good-risk cytogenetic features of t(8;21), t(15;17), or inv 16
      * AML secondary to myelodysplastic disease
  * Acute lymphocytic leukemia (ALL) meeting 1 of the following conditions:

    * In second remission with initial relapse occurring within 2 years of diagnosis
    * In first complete remission with high-risk cytogenetics (t(9;22) or t(4;11))
    * In third or subsequent remission
    * Failed to achieve or sustain a second remission
  * Chronic myelogenous leukemia (CML) in first or second chronic phase or accelerated phase
  * Stage IV lymphoblastic lymphoma not in first remission or that failed to achieve a remission within the first 4 weeks of induction therapy
  * Juvenile CML
  * Myelodysplastic syndrome
  * Severe aplastic anemia unresponsive to anti-thymocyte globulin or cyclosporine
* No CNS or skin involvement with leukemia
* No requirement for mediastinal irradiation
* No healthy, HLA-identical related donor of at least 1 year of age or matched unrelated donor available within 4-6 months
* Availability of a healthy, 1-3 HLA-A, -B, and -DR mismatched related donor

  * Willing and able to undergo general anesthesia for marrow donation and a 5-day course of filgrastim (G-CSF) with 2 daily leukaphereses

PATIENT CHARACTERISTICS:

Age:

* Under 50 (50 and over allowed on a case-by-case basis)

Performance status:

* Age 16 and over:

  * Karnofsky 70-100%
* Under age 16:

  * Lansky 50-100%

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.0 mg/dL (in the absence of liver involvement)
* AST less than twice normal (in the absence of liver involvement)

Renal:

* Creatinine normal OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Asymptomatic or LVEF greater than 50% at rest, with improvement during exercise

Pulmonary:

* Asymptomatic or DLCO greater than 50% predicted (corrected for hemoglobin)

Other:

* No known hypersensitivity to mouse protein or chicken egg products
* No active viral, bacterial, or fungal infection
* HIV-1, HIV-2, HTLV-1, and HTLV-2 negative
* No other concurrent medical condition that would preclude transplantation
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 1995-11; Primary Completion 2004-01 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
overall disease survival | 2 to 4 years post transplant

SECONDARY OUTCOMES:
To correlate progenitor cell doses and doses of clonable T-cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. O'Reilly, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States